CLINICAL TRIAL: NCT00519584
Title: Duration of Interscalene Nerve Blocks With Ropivacaine Alone, Ropivacaine Mixed With Dexamethasone, and Ropivacaine Alone Combined With Systemic Dexamethasone
Brief Title: Interscalene Nerve Blocks With Ropivacaine Alone, With Dexamethasone, Plus Systemic Dexamethasone
Acronym: Ropivacaine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Collected study data was not usable due to process miscommunications
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 07-459
Record Dates: First submitted 2007-08-21; First posted 2007-08-22 (Estimated); Results first posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-06

CONDITIONS: Pain
Keywords: Interscalene nerve block; Dexamethasone; Ropivacaine
MeSH Terms: conditions — Pain | interventions — Ropivacaine; Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ropivacaine/saline (Placebo Comparator): Ropivacaine 30ml 0.5% ropivacaine plus 2 ml 0.9% saline (local placebo) for interscalene block and 0.9% saline 2 ml (systemic placebo) for intravenous injection with sedation for the block
  Interventions: Drug: Ropivacaine; Drug: Saline
- Ropivacaine/dex (Active Comparator): Ropivacaine and local steroid: 30 ml 0.5% ropivacaine plus dexamethasone 8 mg (2 ml) mixed with the local anesthetic and 0.9% saline 2ml (systemic placebo) for intravenous injection with sedation for the block;
  Interventions: Drug: Ropivacaine; Drug: dex
- bupivacaine/dex (Active Comparator): bupivacaine and systemic steroid: 30 ml 0.5% ropivacaine plus 2 ml 0.9% saline (local placebo) for interscalene block plus dexamethasone 8 mg (2 ml) administered intravenously with sedation administered for the block.
  Interventions: Drug: dex; Drug: Bupivacaine
- bupivacaine/Saline (Placebo Comparator): bupivacaine 30ml 0.5% ropivacaine plus 2 ml 0.9% saline (local placebo) for interscalene block and 0.9% saline 2 ml (systemic placebo) for intravenous injection with sedation for the block
  Interventions: Drug: Bupivacaine; Drug: Saline

INTERVENTIONS:
Drug: Ropivacaine — 30 ml 0.5%
  Arms: Ropivacaine/dex; Ropivacaine/saline
Drug: dex — 8 mg (2 ml)
  Other Names: Ropivacaine/dex
  Arms: Ropivacaine/dex; bupivacaine/dex
Drug: Bupivacaine — 30 ml 0.5%
  Arms: bupivacaine/Saline; bupivacaine/dex
Drug: Saline — 0.9% saline; systemic and local
  Other Names: placebo
  Arms: Ropivacaine/saline; bupivacaine/Saline

SUMMARY:
This study will test the hypothesis that ropivacaine in combination with either systemic or local steroid provides comparably longer-lasting analgesia tha ropivacaine alone.

DETAILED DESCRIPTION:
This study proposes to recruit 120 patients who are undergoing open shoulder surgery. Patients will be identified preoperatively by means of the surgical schedule at each participating location. Randomization will be generated by a web-based system and stratified by hospital. The attending physician will be blinded to the contents of the supplied syringes. Treatment assignments consist of three groups:

* Ropivacaine: 30 ml 0.5% ropivacaine plus 2 ml 0.9% saline (local placebo) for interscalene block and 0.9% saline 2 ml (systemic placebo) for intravenous injection with sedation for the block;
* Ropivacaine and local steroid: 30 ml 0.5% ropivacaine plus dexamethasone 8 mg (2 ml) mixed with the local anesthetic and 0.9% saline 2ml (systemic placebo) for intravenous injection with sedation for the block;
* bupivacaine and systemic steroid: 30 ml 0.5% ropivacaine plus 2 ml 0.9% saline (local placebo) for interscalene block plus dexamethasone 8 mg (2 ml) administered intravenously with sedation administered for the block.
* bupivacaine and local steroid: 30 ml 0.5% ropivacaine plus dexamethasone 8 mg (2 ml) mixed with the local anesthetic and 0.9% saline 2ml (systemic placebo) for intravenous injection with sedation for the block;

All solutions for interscalene block will contain epinephrine 1:400,000 as a marker for intravascular injection. Insulated needles with nerve stimulation will be used. Motor response in the surgical limb at a current of < 0.4 mA at 0.1 msec duration will be considered evidence of adequate needle position.

Patients will be evaluated at 5-minute intervals for 15 minutes for development of sensory and motor block. Sensory block will be assessed by loss of sensation to pinprick over the deltoid muscle. Motor block will be assessed by evaluation of ability to abduct the shoulder, the so-called "deltoid sign". During surgery, patients will receive either general anesthesia or sedation at the discretion of the attending anesthesiologist.

Demographic variables, morphometric measurements, and the specific type of procedure will be recorded. The intraoperative management strategy (i.e. general anesthesia versus sedation) and the total doses of fentanyl, midazolam, morphine, and propofol administered perioperatively will be recorded. Finger-stick blood glucose will be measured upon arrival in the postanesthesia care unit (PACU). The primary outcome will be the duration of the interscalene nerve block, which will be measured by time from onset of sensory block until first administration of analgesic medication.

The severity of postoperative pain will be assessed by a blinded observer using a verbal response score (VRS) at 10-minute intervals for 30 minutes in the PACU. Patients reporting pain scores greater than 2 will be given intravenous morphine (1-2 mg) every 5 minutes until they are comfortable. After discharge from the PACU pain unrelieved by oral medication (VRS persistently greater than 4) will be treated with intravenous morphine. Outpatients will receive a prescription for oral acetaminophen with oxycodone.

A blinded observer will interview patients each morning for three days postoperatively. Data collected will include time of block duration,the primary outcome; defined as time from onset of sensory blockade to first administration of supplemental analgesic medication after PACU discharge, as well as secondary outcomes: time to a significant increase in shoulder discomfort, time to a noticeable decrease in numbness and/or weakness, maximum VRS with rest and movement, and total opioid consumption.

The times and VRS scores for secondary outcomes will be based on patient reporting of the corresponding events daily. A member of the study staff will contact patients at 14 days postoperatively to assess for any late or persistent complications such as residual sensory or motor block.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing open shoulder procedures such as rotator cuff repair, capsular shift, subacromial decompression
* Age between 18 and 70 years

Exclusion Criteria:

* Contradictions for interscalene block
* Coagulopathy
* Infection at the needle insertion site
* Moderate to severe chronic obstructive pulmonary disease (COPD)
* Contralateral pneumothorax of diaphragmatic paralysis
* Pregnancy
* Preexisting neuropathy involving the surgical limb
* Systemic glucocorticoid treatment within the last six months of surgery
* Routine opioid use

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2007-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Cummings III, M.D., Principal Investigator — Cleveland Clinic/Hillcrest; Daniel I Sessler, MD, Study Director — The Cleveland Clinic
Locations (2):
- United States (2):
  - Cleveland Clinic Hillcrest, Cleveland, Ohio
  - Cleveland Clinic /Euclid Hospital, Euclid, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ropivacaine/Saline | Ropivacaine/Dex | Bupivacaine/Dex | Bupivacaine/Saline
Started | 54 | 54 | 54 | 56
Completed | 54 | 54 | 54 | 56
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ropivacaine/Saline | Ropivacaine/Dex | Bupivacaine/Dex | Bupivacaine/Saline | Total
Number analyzed (Participants) | 54 | 54 | 54 | 56 | 218
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55 [44 to 55] | 59 [49 to 68] | 58 [53 to 64] | 60 [51 to 68] | 59 [50 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 21 | 19 | 82
  Male | 33 | 33 | 33 | 37 | 136

OUTCOME MEASURES:

1. Primary Outcome: the Duration of Analgesia
Description: the interval between the onset of sensory block and the initial PACU use of opioid analgesia for surgical site pain
Time Frame: surgical date to postoperative day 1 (pod 0 -1 day)
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Ropivacaine/Saline | Ropivacaine/Dex | Bupivacaine/Dex | Bupivacaine/Saline
Number analyzed (Participants) | 54 | 54 | 54 | 56
hours | 22.2 [18 to 28.6] | 11.8 [9.7 to 13.8] | 14.8 [11.8 to 18.1] | 22.4 [20.5 to 29.3]
Statistical Analysis 1: Comparison: Ropivacaine/Saline vs Ropivacaine/Dex; Test type: Superiority; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.17, 95% CI 2-sided [0.08 to 0.39] — Ropivacaine/dex vs. Ropivacaine/saline
Statistical Analysis 2: Comparison: Bupivacaine/Dex vs Bupivacaine/Saline; Test type: Superiority; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.44, 95% CI 2-sided [0.23 to 0.83] — bupivacaine/dex vs. bupivacaine/Saline

2. Secondary Outcome: Time to a Significant Increase in Shoulder Discomfort
Description: the length of time until the patients' first report of surgical site pain.
Time Frame: during postoperative day 1 to 3
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Ropivacaine/Saline | Ropivacaine/Dex | Bupivacaine/Dex | Bupivacaine/Saline
Number analyzed (Participants) | 54 | 54 | 54 | 56
hours | 22.3 [18 to 27.2] | 11.9 [9.2 to 13.8] | 14.7 [13.4 to 17.9] | 25.7 [21.7 to 29.2]
Statistical Analysis 1: Comparison: Bupivacaine/Dex vs Bupivacaine/Saline; Test type: Superiority; p < 0.001, Log Rank
Statistical Analysis 2: Comparison: Ropivacaine/Saline vs Ropivacaine/Dex; Test type: Superiority; p < 0.001, Log Rank

3. Secondary Outcome: Maximum VRS Pain Scores at Rest
Description: Verbal rating scales (VRS): a list of adjectives describing different levels of pain intensity with 0 = no pian and 10 = extremely intense pain. An adequate VRS of pain intensity should include adjectives that reflect the extremes of this dimension; from 'no pain' to 'extremely intense pain'. Patients are asked to read over the list of adjectives and select the word or phrase that best describes their level of pain on the scale from 0 to 10.
Time Frame: postoperative day 1 day 2, day 3.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Ropivacaine/Saline | Ropivacaine/Dex | Bupivacaine/Dex | Bupivacaine/Saline
Number analyzed (Participants) | 54 | 54 | 54 | 56
units on a scale
  POD#1 | 5 [3 to 6.8] | 3.9 [2 to 5.9] | 3 [0 to 4.9] | 4.9 [3 to 7.4]
  POD#2 | 3 [1.9 to 4.2] | 3 [1.9 to 4.8] | 4.1 [3 to 5.9] | 4.1 [2.1 to 4.9]
  POD#3 | 1.9 [0.8 to 3.8] | 2.9 [1.8 to 4.9] | 4 [1.9 to 4.9] | 1.8 [1.1 to 3.8]
Statistical Analysis 1: Comparison: Bupivacaine/Dex vs Bupivacaine/Saline; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — adjusted significance level is 0.025
Statistical Analysis 2: Comparison: Ropivacaine/Saline vs Ropivacaine/Dex; Test type: Superiority; p = 0.005, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Total Opioid Consumption
Description: cumulative opioid consumption in oral oxycodone equivalents (mg) during the first 3 days after surgery.
Time Frame: during first 3 days after surgery
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Ropivacaine/Saline | Ropivacaine/Dex | Bupivacaine/Dex | Bupivacaine/Saline
Number analyzed (Participants) | 54 | 54 | 54 | 56
mg | 75 [45.2 to 152.5] | 79 [45.2 to 100] | 60 [46.7 to 105.2] | 85 [51.3 to 117.6]
Statistical Analysis 1: Comparison: Ropivacaine/Saline vs Ropivacaine/Dex; Test type: Superiority; p = 0.29, Wilcoxon (Mann-Whitney) — adjusted significance level = 0.025
Statistical Analysis 2: Comparison: Bupivacaine/Dex vs Bupivacaine/Saline; Test type: Superiority; p = 0.15, Wilcoxon (Mann-Whitney) — adjusted significance level = 0.025

ADVERSE EVENTS:
Time Frame: after surgery to hospital discharge
Arm/Group | Ropivacaine/Saline | Ropivacaine/Dex | Bupivacaine/Dex | Bupivacaine/Saline
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/54 | 0/54 | 0/56
Other Adverse Events (participants affected / at risk) | 0/54 | 0/54 | 0/54 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No